CLINICAL TRIAL: NCT05066386
Title: Improving the Accuracy of Revised Cardiac Risk Index With HbA1C:Hemoglobin Ratio (HH Ratio)
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H-HHRatio-RCRI
Record Dates: First submitted 2021-09-20; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Risk Stratification; Perioperative Medicine
Keywords: HbA1C: Hemoglobin ratio (HH ratio); Risk model; RCRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Modified RCRI risk stratification — The objective of the study is to compare the predictive value of RCRI and substitution of the "DM on insulin" component with HH ratio for 30- and 90-day mortality, and postoperative acute myocardial injury(AMI) and acute kidney injury(AKI).

SUMMARY:
Retrospective observational study on the effects of altering components of RCRI to improve the predictive capacity.

DETAILED DESCRIPTION:
The current Lee's Revised cardiac risk index (RCRI) was created in 1999. Validation studies have found RCRI to be only moderately discriminant. The "Diabetes Mellitus on insulin" component of the score does not accurately reflect the severity of the disease. A previously studied HbA1C:Hemoglobin ratio shows an improved association with outcomes than individual components alone and could be potentially used as a new marker for severity of the disease.

A retrospective cohort study was performed in consecutive diabetic patients undergoing non-cardiac surgery. Ethics approval was obtained. The objective of the study is to compare the predictive value of RCRI and substitution of the "DM on insulin" component with HH ratio for 30- and 90-day mortality, and postoperative acute myocardial injury(AMI) and acute kidney injury(AKI).

ELIGIBILITY:
* Above 18 years old
* Past medical history of Diabetes Mellitus or preoperative HbA1C > 6.5% (within 3 months of surgery)
* Had HbA1C done within 3 months prior to date of surgery
* Undergoing non cardiac surgery
* Emergency and elective surgery

EXCLUSION:

* If patient is below 18 years old
* no History of DM
* No HbA1C done within 3 months prior to date of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing non cardiac surgery in Singapore General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20099 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 90 days
  To compare the predictive value of RCRI and substitution of the "DM on insulin" component with HH ratio for 30- and 90-day mortality

SECONDARY OUTCOMES:
Morbidity | 7 days
  To compare the predictive value of RCRI and substitution of the "DM on insulin" component with HH ratio for postoperative acute myocardial injury(AMI) and acute kidney injury(AKI).

IPD SHARING:
Plan to Share IPD: No
Due to patient identifiers present in the dataset. Sensitive dataset